CLINICAL TRIAL: NCT03896490
Title: A Feasibility Study of the Attention Control Training (ACT) Intervention Among Very Preterm (VP) Infants
Brief Title: Attention Control Training (ACT) and Very Preterm Infants
Acronym: ACT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Queen's University, Belfast (Other)
Collaborators: Public Health Agency, Health and Social Care Research and Development (Other); TinyLife (Other)
Responsible Party: Principal Investigator, Oliver Perra, Principal Investigator, Queen's University, Belfast
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: R4798NUR
Record Dates: First submitted 2019-03-27; First posted 2019-04-01 (Actual); Results first posted 2023-07-25 (Actual); Last update posted 2023-07-25 (Actual); Status verified 2022-09

CONDITIONS: Very Premature Baby
Keywords: Learning; Memory; Memory Training; Attention; Computerized Cognitive Training

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ACT (Experimental)
  Interventions: Behavioral: Attention Control Training
- Control (Placebo Comparator)
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: Attention Control Training — Infants watch interactive cartoons that respond to infants' direction of gaze. An eye-tracker records the infant's eye movements in real time, relaying this information to the computer. These presentations trigger motivating stimuli (cartoon animations with child-friendly sounds) every time the infant fulfills the demands of a task (e.g. when the infant looks at a character on the screen avoiding to be distracted by other objects moving across the screen). The length of training sessions varies depending on infants' engagement with stimuli and time criteria.
  Arms: ACT
Behavioral: Control — The control procedure involves presentation of cartoons on a screen, while infants' gaze direction is recorded using the same eye-tracker and camera. The crucial difference is that the cartoons in this case are not interactive, thus do not change depending on infants' gaze direction. To ensure presentations in the control procedure are similar in length to those of the intervention group, infants in the control group are matched infant-by-infant and visit-by-visit with participants in the ACT treatment group: Infants in the control group see a replay of the session of the matched treated infant. Therefore, while the presentation is exactly the same (i.e. same length and same stimuli) for the treated and the control child, in the latter case the presentation is not interactive (i.e. not generated contingently on the infants' visual behaviour).
  Arms: Control

SUMMARY:
Infants' attention control, defined as the ability to select what to pay attention to, is a fundamental building block for developing learning abilities and behaviour self-regulation. Infants born before term (<37 weeks gestation) display delays in attention control, and these delays cause cascade effects that include learning difficulties and behaviour problems. Infants born before 32 weeks of gestation, known as very preterm (VP), are particularly at risk of persistent difficulties in attention.

A ground-breaking early intervention, the Attention Control Training (ACT), targets infants' attention control. The novelty of the ACT lies in engaging young infants in "brain-training" using a computer interface, which tracks infants' gaze direction and presents training visual stimuli appropriate to the infants' ability level. Results demonstrate ACT improves attention of typically developing infants, contributing to improvements in other cognitive abilities (e.g. memory), but ACT has not been tested in clinical populations such as VP infants.

The investigators are running a feasibility study of the ACT intervention amongst VP infants aged 1 year (corrected age for prematurity). This feasibility study is necessary in order to adapt the ACT material and presentation to VP infants, and in particular to investigate the acceptability of a Randomised Trial and its training schedule by parents of VP infants.

The proposed study will allow the investigators to identify solutions to problems, ensuring the ACT material and delivery are customised for VP infants.

DETAILED DESCRIPTION:
The aims of this project are to:

1. Investigate VP infants' engagement with the ACT procedure;
2. Assess the quality of data collected during the training and assessments used, and compare them to similar data obtained from typically developing infants who completed studies conducted by collaborators.
3. Investigate retention into the programme.
4. Investigate infants' performance in outcome measures and assess trends indicating differences in performance between treated and controls.

To allow for a fair test of the ACT, infants will be randomly assigned to receive the ACT programme or to watch age appropriate non-interactive cartoons (control procedure). By randomly assigning infants to the ACT or the control procedure, the investigators can be sure that infants in the treatment group do not differ systematically from those in the control group: the two groups will therefore differ only for effect of chance, and the only systematic difference between them will lie in the experimental treatment.

All the assessments will take place in a dedicated room. The use of a dedicated room will ensure that infants are assessed in controlled conditions whereby interference from noise, changes in light, or other sources of distraction, are minimised.

The first session will take place by the time the infant is aged 12 months (age corrected for prematurity). This session will include a baseline assessment followed by a first training/control procedure (depending on the child's random assignment in one group or the other). During the baseline assessment parents will be asked to answer questions about the family and infants' behaviour.

The investigators will also assess infants' attention using computer-based tasks whereby infants have to watch some images on a screen (e.g. pictures of babies, cartoon characters, etc.), as well as using tasks whereby infants are asked to play with novel toys or interact with the researcher. The investigators will also collect a general assessment of the infants' cognitive skills using the Mullen scales, a validated and age-appropriate battery. Finally, the investigators will record mother and infant playing together for some minutes in order to assess infants' abilities to pay attention and focus on other people and objects in a naturalistic situation, similar to familiar play routines at home.

After the assessment, the researcher tasked with running the ACT or control procedure will open a sealed envelope and will find out to which group (ACT or control) the child has been assigned. If the infant is still in an alert and attentive state, the experimenter will proceed with the delivery of the ACT or control procedure accordingly to the infant's assignment.

Parents will not be told what type of videos (ACT or control) their child will be watching. This is to ensure that parents do not change their behaviour when they know to which procedure their child is taking part. The cartoons displayed to the control group will be identical to those shown to the treated: the only (pivotal) difference will lie in that the cartoons will be interactive (i.e. activated contingently on infant's gaze behaviour) for the treated, while they will not be interactive for infants in the control group. Since the cartoons will be identical across groups, and, furthermore, parents will not be able to detect the direction of gaze of the infant during training while infants are held on the parent's lap, the investigators believe that it will be difficult for parents to recognise their infant's group allocation. However, the research team will investigate this by asking a series of follow-up questions to parents at the end of the study.

Infants will be allocated to one of two groups :

1. the ACT training programme delivered across 4 consecutive weekly sessions for a month (n=10);
2. Control (n=10), whereby infants will be shown cartoons over the same number of weekly sessions and for a corresponding amount of time as infants in the ACT intervention.

Weekly session 2, 3, and 4 will involve further administration of training/control procedures.

The final session in week 5 will involve collection of outcome measures. The same questionnaires and tasks described in the baseline assessment will be used. The researcher that will assess the infant in the 5th session will be a blind assessor (who will not know in which group, ACT or Control, the infant has been allocated).

ELIGIBILITY:
Inclusion Criteria:

* Infants born very preterm (gestational age 28 to less than 32 weeks);
* Infant's family residing in Northern Ireland;
* Infant's age 12 months (+/- 1 month) at the start of the study, corrected for prematurity

Exclusion Criteria:

* Significant visual and/or hearing disabilities;
* Congenital anomalies that may impact on their cognitive and sensory-motor development;
* A diagnosis of Cerebral Palsy;
* Infant taking part in a trial (or have recently taken part in a trial) which may interfere with this study (e.g. by affecting concentration abilities or representing a significant burden for the family).

Ages: 11 Months to 13 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 12 (Actual)
Dates: Start 2018-03-11 (Actual); Primary Completion 2019-06-28 (Actual); Study Completion 2020-03-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Queen's University Belfast, Belfast, Northern Ireland, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Perra O, Wass S, McNulty A, Sweet D, Papageorgiou K, Johnston M, Patterson A, Bilello D, Alderdice F. Training attention control of very preterm infants: protocol for a feasibility study of the Attention Control Training (ACT). Pilot Feasibility Stud. 2020 Feb 10;6:17. doi: 10.1186/s40814-020-0556-9. eCollection 2020. PMID 32055404
- [Derived] Perra O, Alderdice F, Sweet D, McNulty A, Johnston M, Bilello D, Papageorgiou K, Wass S. Attention and social communication skills of very preterm infants after training attention control: Bayesian analyses of a feasibility study. PLoS One. 2022 Sep 22;17(9):e0273767. doi: 10.1371/journal.pone.0273767. eCollection 2022. PMID 36137090
- [Derived] Perra O, Wass S, McNulty A, Sweet D, Papageorgiou KA, Johnston M, Bilello D, Patterson A, Alderdice F. Very preterm infants engage in an intervention to train their control of attention: results from the feasibility study of the Attention Control Training (ACT) randomised trial. Pilot Feasibility Stud. 2021 Mar 12;7(1):66. doi: 10.1186/s40814-021-00809-z. PMID 33712090
- See also: Paper describing the study protocol — https://doi.org/10.1186/s40814-020-0556-9

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The recruitment phase encompassed 13 months from April 2018 to April 2019. Eligible participants were identified by two categories of gatekeepers: (a) Collaborating neonatology practitioners in hospitals within the Belfast, South Eastern, and Northern Trust in Northern Ireland; (b) A local charity for families of premature children. The gatekeepers ensured that parents or caregivers of eligible infants received information about the study.
Groups:
- Attention Control Training: ACT: Infants watch interactive cartoons that respond to infants' direction of gaze. An eye-tracker records the infant's eye movements in real time, relaying this information to the computer. These presentations trigger motivating stimulations (cartoon animations with child-friendly sounds) every time the infant fulfills the demands of a task (e.g. when the infant looks at a character on the screen avoiding to be distracted by other objects moving across the screen). The length of training sessions varies depending on infants' engagement with stimuli and time criteria.
- Control: Control: The control procedure involve presentation of cartoons on a screen, while infants' gaze direction will also be recorded using the same eye-tracker and camera. The crucial difference is that the cartoons in this case are not interactive, thus do not change depending on infants' gaze direction. To ensure presentations in the control procedure are similar in length to those of the intervention group, infants in the control group are matched infant-by-infant and visit-by-visit with participants in the ACT treatment group: Infants in the control group see a replay of the session of the matched treated infant. Therefore, while the presentation is exactly the same (i.e. same length and same stimuli) for the treated and the control child, in the latter case the presentation is not interactive (i.e. not generated contingently on the infants' visual behaviour).
Period: Overall Study
Arm/Group | Attention Control Training | Control
Started | 6 | 6
Completed | 5 | 5
Not Completed | 1 | 1
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Population: Participants randomly allocated to the two arms. The random allocation sequence was created in two blocks (n=10 each) using randomly-generated numbers from the uniform distribution. The intervention/control ratio was constrained to be 1:1.
Groups:
- Attention Control Training: ACT: Infants watch interactive cartoons that respond to infants' direction of gaze. An eye-tracker records the infant's eye movements in real time, relaying this information to the computer. These presentation trigger motivating stimulations (cartoon animations with child-friendly sounds) every time the infant fulfils the demands of a task (e.g. when the infant looks at a character on the screen avoiding to be distracted by other objects moving across the screen). The length of training sessions varies depending on infants' engagement with stimuli and time criteria.
- Control: Control: The control procedure will involve presentation of cartoons on a screen, while infants' gaze direction will also be recorded using the same eye-tracker and camera. The crucial difference will be that the cartoons in this case are not interactive, thus do not change depending on infants' gaze direction. To ensure presentations in the control procedure are similar in length to those of the intervention group, infants in the control group will be matched infant-by-infant and visit-by-visit with participants in the ACT treatment group: Infants in the control group will see a replay of the session of the matched treated infant. Therefore, while the presentation will be exactly the same (i.e. same length and same stimuli) for the treated and the control child, in the latter case the presentation will not be interactive (i.e. not generated contingently on the infants' visual behaviour).
- Total: Total of all reporting groups
Arm/Group | Attention Control Training | Control | Total
Number analyzed (Participants) | 6 | 6 | 12
Age, Continuous [Mean (Standard Deviation); unit: Months (Corrected Age)] — Population: One participant did not attend the pre-test session (withdrew before starting the study)
  Months (Corrected Age)
    number analyzed (Participants) | 5 | 6 | 11
    (all) | 11.90 (0.79) | 13.04 (1.21) | 12.52 (1.16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 4 | 4 | 8
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United Kingdom | 6 | 6 | 12
Gestational Age [Mean (Standard Deviation); unit: Weeks] — Population: One participant did not attend the pre-test session
  Weeks
    number analyzed (Participants) | 5 | 6 | 11
    (all) | 29.20 (1.09) | 30.00 (1.09) | 29.64 (1.12)
Birth Weight [Mean (Standard Deviation); unit: grams] — Population: One participant did not attend the pre-test session
  grams
    number analyzed (Participants) | 5 | 6 | 11
    (all) | 1313 (338) | 1378 (332) | 1349 (319)
Main caregiver's highest educational attainment [Count of Participants; unit: Participants] — Population: One participant in the Intervention arm did not attend the pre-test, therefore information was not collected. A participant in the control arm did not provide the information
  Participants
    number analyzed (Participants) | 5 | 5 | 10
    University Degree or higher | 5 | 3 | 8
    Other | 0 | 2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Recruitment and Retention
Description: Recruitment as a percentage of the eligible families approached who agreed to take part in the study and were randomised, and retention, defined as the percentage of randomised participants for whom data are available at baseline and post-test.
Time Frame: 1 year
Population: Overall, of all the families eligible and contacted by the gatekeepers, 27 recorded their interest for the study by contacting the research group: Seven of these families had twins, thus representing 34 eligible participants that expressed interest in the study. Out of these, 11 families agreed to take part (41% of those who recorded their interest). These accounted for 12 infants being randomised to take part in the study, as one family had twins.
Measure: Count of Participants; unit: Participants
Groups:
- Attention Control Training: ACT: Infants watch interactive cartoons that respond to infants' direction of gaze. An eye-tracker records the infant's eye movements in real time, relaying this information to the computer. These presentations trigger motivating stimuli (cartoon animations with child-friendly sounds) every time the infant fulfills the demands of a task (e.g. when the infant looks at a character on the screen avoiding to be distracted by other objects moving across the screen). The length of training sessions varies depending on infants' engagement with stimuli and time criteria.
Arm/Group | Attention Control Training | Control
Number analyzed (Participants) | 6 | 6
Participants | 5 | 5

2. Secondary Outcome: Percentage of Training/Control Sessions Attended by Infants
Description: Sessions attended are defined as sessions to which parent and infant are present at the scheduled appointment
Time Frame: 1 year
Population: Percentage of sessions attended by infants
Measure: Mean (Standard Deviation); unit: percentage of visits attended
Arm/Group | Attention Control Training | Control
Number analyzed (Participants) | 5 | 5
percentage of visits attended | 100 (0) | 100 (0)

3. Secondary Outcome: Percentage of Training/Control Sessions Completed by Infants
Description: Sessions completed are defined as sessions whereby infants engaged without interruptions for at least 240 sec in at least two tasks.
Time Frame: 1 year
Population: Percentages of tasks completed by infants in the two arms in each session
Measure: Mean (Standard Deviation); unit: percentage of tasks completed
Arm/Group | Attention Control Training | Control
Number analyzed (Participants) | 5 | 5
percentage of tasks completed | 73.16 (26.63) | 72.92 (24.26)

4. Secondary Outcome: Duration of Tasks Administered to Infants During Training/Control Sessions
Description: Duration is defined as the cumulative duration in seconds of the tasks delivered to infants during the training or control sessions.
Time Frame: 1 year
Population: Cumulative duration of tasks completed
Measure: Mean (Full Range); unit: minutes
Arm/Group | Attention Control Training | Control
Number analyzed (Participants) | 5 | 5
minutes | 83.60 [65.95 to 104.05] | 75.07 [61.41 to 87.88]

5. Secondary Outcome: Percentage of Tasks Completed at Post-test
Description: Completion is defined according to time criteria specific for each of the four attention tasks. Specifically, a sustained attention stipulates an infant completes two consecutive looks at less than 50% of the longest look displayed, or 120 s of accumulated looking time, or 12 trials without showing consecutive looks at less than 50% of the longest look displayed (habituation criterion). A visual-paired comparison task stipulates that stimuli are displayed for 16,000 ms. A disengagement task stipulates administration of at least 52 trials. An information density preference task stipulates administration of 6 blocks of the task in total.
Time Frame: 1 year
Population: Percentage of tasks completed during post-test
Measure: Mean (Standard Deviation); unit: percentage of tasks completed
Arm/Group | Attention Control Training | Control
Number analyzed (Participants) | 6 | 6
percentage of tasks completed | 80.95 (39.50) | 80.95 (39.50)

6. Secondary Outcome: Quality of Eye-tracker Data Collected During Baseline and Post-test Attention Assessments
Description: A random sample of the baseline and post-test attention assessments will be selected at random (20% of all the completed assessments). The quality of the eye-tracker data collected will be assessed by determining the number of usable fragments recorded during the task and the proportion of usable fragments recorded by the duration of the task in seconds.
Time Frame: 1 year
Population: Flicker was defined as the duration in seconds of usable fragments of eye-tracking data during the task recording. The loss of usable fragments during a recording can be caused by unavailability of any of the elements the eye-tracker uses to assess gaze direction (e.g. when infants turn away from the screen). Thus, a longer duration indicated more robust recordings.
Measure: Mean (Standard Error); unit: seconds
Arm/Group | Attention Control Training | Control
Number analyzed (Participants) | 5 | 5
seconds | 1.84 (1.39) | 1.21 (0.68)

7. Secondary Outcome: Performance During Training
Description: Performance indicators included reaction times or level of task difficulty achieved. These indicators were standardized (std.): higher scores indicated better performance and followed a normal distribution with ranges roughly between -3 and +3. Each infant contributed several performance scores during each visit. We used multilevel growth regression models to test if trained infants displayed linear changes in performance across visits: linear effects would indicate significant performance improvement across tasks. In these analyses, the units of observations were the std. scores registered across visits, which were considered nested within infants. The models allowed to estimate the initial status (average std. scores in the first visit) and the rate of change (the average change in performance std. scores from one visit to another), as well as residual variances around these parameters
Time Frame: 1 year
Population: We report infants' rate of change across the Target Search tasks. This information was meaningful only in the Intervention group, insofar searching for targets on the screen determined the interactive displays on the screen to change accordingly. In the control group these displays followed a pre-set schedule (non-interactive displays) therefore the infants' behaviour had no effect on the display, and was thus not measured.
Measure: Mean (95% Confidence Interval); unit: standardised scores
Arm/Group | Attention Control Training | Control
Number analyzed (Participants) | 5 | 0
standardised scores | 0.40 [0.04 to 0.76] |

ADVERSE EVENTS:
Time Frame: 18 months
Description: Any untoward or unfavorable medical occurrence in a participant, including any abnormal sign (for example, abnormal physical exam or laboratory finding), symptom, or disease, temporally associated with the participant's participation in the research, whether or not considered related to the participant's participation in the research.
Arm/Group | Attention Control Training | Control
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 0/6 | 0/6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-11-16): https://cdn.clinicaltrials.gov/large-docs/90/NCT03896490/Prot_SAP_000.pdf